CLINICAL TRIAL: NCT04192526
Title: Assessment of Serum Cholinesrtrase Level in Aluminum Phosphide Poisoning Cases, the Possible Proposing Role of Atropine and Pralidoxime in Saving the Cases: Clinical and
Brief Title: Serum Cholinesterase Level in Aluminum Phosphide Poisoning, the Possible Proposing Role of Atropin & Pralidoxime
Acronym: ALPH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Abd El-Rahman, lecture, Assiut University
Other Study IDs: serum cholinestrase in AP
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Toxicity;Chemical
Keywords: serum cholinestrase, atropin, aluminum phosphide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metal phosphides are widely used as a rodenticide and insecticide and poisoning with these substances has a very high mortality. The aim of this study was to evaluate the butyrylcholinesterase (BuCh) level in poisoning with metal phosphides.

DETAILED DESCRIPTION:
Today, the use of pesticides in the world is considered as a recognized health It is estimated that around 30% of global suicides are due to pesticide self-poisoning . Metal phosphides pesticides are highly toxic, low cost, and are easily accessible as rodenticide agents and used for self-poisoning . aluminum phosphide (ALP) are among the most important metal phosphides. Poisoning with these agents is frequently seen in India, Srilanka and Iran. In a recent study, the incidence of fatal aluminum phosphide poisoning cases referred for phosphine analysis was 5.22 and 37.02 per million of population of Tehran, Iran in 2006 and 2013, respectively (9).The mechanism of toxicity is not clearly defined. ALP toxicity is related to the production of phosphine gas. Phosphine inhibits cytochrome c oxidase and causes mitochondrial destruction and inhibits oxidative respiration which leads to anaerobic metabolism, severe metabolic acidosis, multi-organ dysfunction and death. Phosphine can lead to severe cardiac suppression and cardiogenic shock. One of the proposed mechanisms of toxicity is the reduction of the true cholinesterase and serum cholinesterase (butyrylcholinesterase) enzyme, but usually do not show obvious clinical manifestations .

ELIGIBILITY:
Inclusion Criteria: cases of aluminum phosphide poisoning -

Exclusion Criteria: concomitant ingestion

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cases of aluminum phosphide poisoning attending Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
persistent cholineastrase inhibition is one of the pathological pathway of the ALP poisoning | 3 months
  definite assessment of the pathogenesis of ALP helps in applying adaquqte treatment regmin

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Abd el rahman, Principal Investigator — AssiutU, faculty of medicine
Locations (1):
- AssiutU, Asyut, Egypt